CLINICAL TRIAL: NCT06680310
Title: Prospective Multicenter Study of Ultrasound Evaluation of Salivary Glands in Patients with Sjögren's Disease Compared with Patients with Connective Tissue Diseases (lupus, Scleroderma, Rheumatoid Arthritis) and Healthy Subjects with Dry Syndromes
Brief Title: Ultrasonic COmparison of Salivary Glands in Autoimmune Diseases (COUGAR)
Acronym: COUGAR
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Collaborators: CHRU de Brest (Brest University Hospital) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0273; 2024-A00412-45 (Other: ANSM)
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Sjogren Syndrome; Dry Syndrome; Lupus; Scleroderma; Rheumatoid Arthritis
MeSH Terms: conditions — Sjogren's Syndrome; Scleroderma, Diffuse; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Sjogren syndrome: Ultrasound of the parotid and submandibular salivary glands in routine care of patients with Sjögren
- Other autoimmune diseases (Lupus/RA/Scleroderma): Ultrasound of the parotid and submandibular salivary glands in routine care of patients with other autoimmune diseases (Lupus/RA/Scleroderma)
- Dry syndrome: Ultrasound of the parotid and submandibular salivary glands in routine care of patients with dry syndrome

SUMMARY:
Prospective multicenter cross-sectional study evaluating ultrasound of the main salivary glands (2 parotid and 2 submandibular) in patients with Sjögren's disease compared with patients with other connective diseases (rheumatoid arthritis (RA), lupus, scleroderma) and control patients (patient with dry syndrome without the above-mentioned autoimmune disease).

DETAILED DESCRIPTION:
This is a non-interventional study involving patients who are routinely monitored for their disease, and who typically benefit from ultrasound of the parotid and submandibular salivary glands as part of their dry mouth syndrome. Recruitment will be facilitated by the fact that these will be "general population" patients with Sjögren's disease, lupus, RA, scleroderma with dry syndrome, and control patient.

The study will be conducted over a single visit, including a clinical examination and an ultrasound scan. Ultrasound will not be blinded to the clinic, so we will need only one examiner per center.

This is a study in routine care, with no additional costs and no expected constraints. The examination will be carried out as part of their routine follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Patients fulfilling Sjogren criteria (2012 and 2016 American-European criteria) or Lupus according to ACR 2019 criteria or RA according to ACR/EULAR 2010 criteria or scleroderma according to ACR-EULAR 2013 classification criteria or control patient (patient with dry syndrome felt without pre-cited autoimmune disease).

Exclusion Criteria:

* Uncooperative patient who has refused to participate in the study.
* Patients unable to understand the protocol, under guardianship or curatorship.
* Patients not affiliated to the French Social Security system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Sjögren's disease, all patients with autoimmune diseases such as LUPUS, scleroderma or rheumatoid arthritis with dry syndrome, and a population of healthy controls with dry syndrome and no autoimmune disease as mentioned above.
Sampling Method: Non-Probability Sample
Enrollment: 501 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the rate of patients with structural anomalies of the salivary glands, for each of three populations | Baseline
  The salivary gland assessment score will be evaluated according to the OMERACT score (0-3) for each group of patients.

SECONDARY OUTCOMES:
Evaluate the proportion of patients with ultrasound abnormalities in each subgroup. | Baseline
  Evaluate the proportion of patients with B-mode ultrasound abnormalities (0-3) in each subgroup.
Evaluate the proportion of patients with vascular anomalies in each subgroup | Baseline
  Study of the contribution of Doppler ultrasound to the study of salivary gland vascularization in each subgroup

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: No